CLINICAL TRIAL: NCT01301729
Title: A Multicenter, Single Arm, Open-Label PhIV Study to Investigate the Effect of First-Line Herceptin (Trastuzumab) in Combination With a Taxane in Patients With Metastatic Breast Cancer Who Relapsed After Receiving (Neo)Adjuvant Herceptin for HER2-Positive Early Breast Cancer
Brief Title: A Study of Herceptin (Trastuzumab) in Combination With a Taxane in Participants With HER2-Positive Breast Cancer Who Relapsed After (Neo)Adjuvant Herceptin Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25288
Record Dates: First submitted 2011-02-09; First posted 2011-02-23 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Paclitaxel; Trastuzumab

ARMS (1):
- Trastuzumab (Experimental): Participants with metastatic breast cancer received a loading dose of 4 milligrams per kilograms (mg/kg) of trastuzumab intravenously (IV) followed by 2 mg/kg of trastuzumab IV once a week along with docetaxel 100 milligrams per meter square (mg/m^2), every 3 weeks or paclitaxel 90 mg/m^2 once a week until progression of disease, occurrence of intolerable toxicity, the participant discontinues the study or dies.
  Interventions: Drug: Docetaxel; Drug: Paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Docetaxel — 100 mg/m2 iv every 3 weeks, 6 cycles (18 weeks)
Drug: Paclitaxel — 90 mg/kg iv (+/-10%) every 3 weeks for 6 3-week cycles (18 weeks)
Drug: Trastuzumab — 4 mg/kg iv loading dose on Day 1, 2 mg/kg iv on Day 8 and weekly thereafter
  Other Names: Herceptin

SUMMARY:
This single arm, open-label study will evaluate the efficacy and safety of Herceptin (trastuzumab) in combination with a taxane as first line therapy in participants with HER2-positive breast cancer who relapsed after neoadjuvant or adjuvant Herceptin treatment. Participants will receive Herceptin (loading dose of 4 mg/kg intravenously [iv], 2 mg/kg iv weekly thereafter) with 6 3-week cycles of either docetaxel (100 mg/m2 iv every 3 weeks) or paclitaxel (90 mg/m2 every week). Herceptin treatment will be continued until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Female participants , >/= 18 years of age
* Locally recurrent/metastatic breast cancer (relapse in supra- or infraclavicular lymph nodes is regarded as metastatic disease)
* HER2-positive primary disease
* Participants must have received Herceptin in the adjuvant and/or neoadjuvant setting
* Relapsed breast cancer >/= 6 months after discontinuing last drugs of Herceptin and/or chemotherapy in the adjuvant and/or neoadjuvant setting for HER2-positive breast cancer
* Measurable disease according to RECIST 1.0
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Maximum cumulative dose of doxorubicin </= 360 mg/m2 or of epirubicin </= 720 mg/m2 or no prior anthracyclines
* At least 3 weeks after prior surgery or radiotherapy

Exclusion Criteria:

* Pregnant or breastfeeding women
* Previous chemotherapy for metastatic breast cancer (prior endocrine therapy till progressive disease is allowed)
* Pleural effusions, ascites or bone lesions as only manifestation of disease
* Brain metastases
* Invasive malignancy other than metastatic breast cancer
* Inadequate bone marrow, hepatic or renal function
* Prior treatment with anti-HER therapies other than (neo)adjuvant Herceptin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- China (10):
  - Beijing
  - Chengdu
  - Guangzhou
  - Hangzhou
  - Harbin
  - Nanjing
  - Shanghai
  - Shenyang
  - Wuhan
  - Zhengzhou

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 32 participants were enrolled in the study and received study treatment.
Period: Overall Study
Arm/Group | Trastuzumab
Started | 32
Completed | 28
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Participant did not Return for Treatment | 1
Not completed — Violated Selection Criteria | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) data set is defined as all the participants who are eligible through screening, register and enter the study.
Arm/Group | Trastuzumab
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (11.61)
Gender [Count of Participants; unit: Participants]
  Female | 32
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was assessed according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.0 and was defined as the time from the date when the participant signed the informed consent form (ICF) until death or progressive disease (PD). PD was defined as 20% increase in the sum of the longest diameter of target lesions. PFS and associated confidence intervals were calculated using the Kaplan-Meier method.
Time Frame: From the date of informed consent to the date of death or progressive disease (up to 28 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab
Number analyzed (Participants) | 32
months | 9.9 [6.28 to 13.63]

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate was assessed using RECIST 1.0 and defined as the percentage of participants that achieved a complete response (CR) or a partial response (PR). CR was defined as complete disappearance of all target and non-target lesions and no new lesions. PR was defined as greater than or equal to (≥) 30 % decrease in the sum of appropriate diameters of all target measurable lesions, no progress in the non-measurable disease, and no new lesions.
Time Frame: up to 28 months
Population: ITT data set is defined as all the participants who are eligible through screening, register and enter the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tastuzumab: Participants with metastatic breast cancer received a loading dose of 4 milligrams per kilograms (mg/kg) of trastuzumab intravenously (IV) followed by 2 mg/kg of trastuzumab IV once a week along with docetaxel 100 milligrams per meter square (mg/m^2), every 3 weeks or paclitaxel 90 mg/m^2 once a week until progression of disease, occurrence of intolerable toxicity, the participant discontinues the study or dies.
Arm/Group | Tastuzumab
Number analyzed (Participants) | 32
percentage of participants | 81.3 [63.6 to 92.8]

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from when a PR or CR was first documented until the date of documented PD or death. CR was defined as complete disappearance of all target and non-target lesions and no new lesions. PR was defined as greater than or equal to (≥) 30 % decrease in the sum of appropriate diameters of all target measurable lesions, no progress in the non-measurable disease, and no new lesions. PD was defined as 20% increase in the sum of the longest diameter of target lesions.
Time Frame: From the time of PR or CR until the date of PD or death (up to 28 months)
Population: ITT data set is defined as all the participants who are eligible through screening, register and enter the study. Here, number of participants are the participants who had response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab
Number analyzed (Participants) | 26
months | 9.8 [5.82 to 11.60]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of enrollment to the date of death due to any cause.
Time Frame: Time from enrollment to the date of death (up to 28 months)
Population: ITT data set is defined as all the participants who are eligible through screening, register and enter the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab
Number analyzed (Participants) | 32
months | NA [22.64 to NA] — The median for overall survival was not reached as insufficient number of participants had event.

5. Secondary Outcome: Percentage of Participants With an Adverse Event (AE)
Description: An AE was defined as any adverse medical event that occurred after the participant used the investigational medicinal product (IMP) or other intervention behaviors specified by the protocol in the clinical trial regardless of relationship to the study treatment.
Time Frame: Up to 28 days after last infusion of the study drug (28 months)
Population: Safety population is defined as all enrolled participants and have taken at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 32
percentage of participants | 93.8

6. Secondary Outcome: Determination of Biomarkers Indicative for Response (Serum and Tumour Tissue Analyses)
Time Frame: up to 28 months
Population: Biomarker analysis was not performed as the eligible biomarker sample quantity was too limited for testing.
Arm/Group | Trastuzumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate was assessed according to RECIST 1.0 and defined as the percentage of participants who experienced a CR, PR, or stable disease (SD) for at least 6 months. CR was defined as complete disappearance of all target and non-target lesions and no new lesions. PR was defined as greater than or equal to (≥) 30 % decrease in the sum of appropriate diameters of all target measurable lesions, no progress in the non-measurable disease, and no new lesions. SD was defined as small changes that do not meet above criteria.
Time Frame: up to 28 months
Population: ITT data set is defined as all the participants who are eligible through screening, register and enter the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 32
percentage of participants | 81.3 [63.6 to 92.8]

8. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from the date of enrollment until the date of progressive disease.
Time Frame: From the date of enrollment until the date of progressive disease (up to 28 months)
Population: ITT data set is defined as all the participants who are eligible through screening, register and enter the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab
Number analyzed (Participants) | 32
months | 9.9 [6.28 to 13.63]

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last dose of the study drug (up to 28 months)
Description: An AE was defined as any adverse medical event that occurred after the participant used the investigational medicinal product (IMP) or other intervention behaviors specified by the protocol in the clinical trial regardless of relationship to the study treatment.
Arm/Group | Trastuzumab
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=32)
Infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Completed suicide (Psychiatric disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Cataract (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=32)
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Transaminases increased (Investigations) | 2
Hypoaesthesia (Nervous system disorders) | 11
Headache (Nervous system disorders) | 3
Insomnia (Nervous system disorders) | 2
Neurotoxicity (Injury, poisoning and procedural complications) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 3
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 7
Nail disorder (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 3
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 3
Paronychia (Skin and subcutaneous tissue disorders) | 2
Asthenia (General disorders) | 7
Pyrexia (General disorders) | 6
Oedema peripheral (General disorders) | 5
Flushing (General disorders) | 2
Face oedema (General disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 5
Hypophagia (Gastrointestinal disorders) | 5
Vomting (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 19
Neutropenia (Blood and lymphatic system disorders) | 18
Agranulocytosis (Blood and lymphatic system disorders) | 10
Bone marrow failure (Blood and lymphatic system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.